CLINICAL TRIAL: NCT06273891
Title: Erythromycin Versus Azithromycin for Preterm Prelabor Rupture of Membranes: A Cluster Randomized Comparative Effectiveness Trial
Brief Title: Erythromycin Versus Azithromycin for Preterm Prelabor Rupture of Membranes
Acronym: PRACET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INOVA-2023-58; 23-08-WC-0198 (Other: Eastern Virginia Medical School)
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Premature Rupture of Membrane
Keywords: pprom; latency antibiotics; prom
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes | interventions — Erythromycin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erythromycin (Active Comparator): Erythromycin 250 mg IV every 6 hours for 48 hours, followed by 250 mg PO or 333 mg PO every 8 hours for 5 days
  Interventions: Drug: Erythromycin
- Azithromycin (Active Comparator): Azithromycin 1 gm PO once or 500 mg PO followed by 250 mg PO daily for a total of 5 days
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Erythromycin — Erythromycin 250 mg IV every 6 hours for 48 hours, followed by 250 mg PO or 333 mg PO every 8 hours for 5 days
  in addition to Ampicillin 2 gm IV every 6 hours for 2 days followed by Amoxicillin 250 mg PO every 8 hours for 5 days
  Arms: Erythromycin
Drug: Azithromycin — Azithromycin 1 gm PO once or 500 mg PO followed by 250 mg PO daily for a total of 5 days
  in addition to Ampicillin 2 gm IV every 6 hours for 2 days followed by Amoxicillin 250 mg PO every 8 hours for 5 days
  Arms: Azithromycin

SUMMARY:
The goal of this study is to help identify the best antibiotic treatment for pregnant people when their water breaks prematurely (a condition abbreviated as PPROM). Current practice is to attempt to maintain the pregnancy until at least 34 weeks gestational age, when the risks of prematurity to the baby are lessened. Research shows that antibiotics help the pregnancy last longer, but there have been limited studies about which combination works best. Currently, both azithromycin and erythromycin are accepted antibiotic treatments, in addition to ampicillin and amoxicillin. Participants diagnosed with PPROM will be randomized to receive ampicillin and amoxicillin plus either azithromycin or erythromycin, in addition to the care they would normally receive. Studying these two drugs will help decide the best care for future patients with PPROM.

DETAILED DESCRIPTION:
Preterm pre-labor rupture of membranes (PPROM) complicates 3% of pregnancies and accounts for one-fourth to one-third of preterm births. PPROM is associated with significant maternal and neonatal morbidities, including chorioamnionitis, endometritis, neonatal sepsis, prematurity-related pathologies. In the absence of labor or indication for immediate delivery, patients who present at less than 34 weeks gestational age are treated with antibiotics to prolong pregnancy until 34 weeks when the risks of prematurity are decreased. Based on randomized trials, both the American College of Obstetrics and Gynecology (ACOG) and the Society of Maternal Fetal Medicine (SMFM) recommend IV ampicillin and IV erythromycin for 2 days, followed by an oral regimen of amoxicillin and erythromycin for 5 days. Due to the recent limited availability of erythromycin, azithromycin has been used a substitute. There have been observational studies showing no difference in duration of pregnancy between azithromycin and erythromycin, however no randomized controlled trial has been carried out to our knowledge. This study performs a cluster randomized controlled trial to examine the efficacy of azithromycin versus erythromycin as a component of the "latency antibiotics" used to prolong pregnancy in PPROM patients.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy at 22 weeks 0 days to 32 weeks 6 days of gestation.
* Rupture of membranes confirmed by biochemical testing.
* Membrane rupture within the past 36 hours.
* Cervical dilation 3 cm or less and 4 or fewer contractions within 60-minutes at the time of admission.
* Age ≥18 and <50 years.

Exclusion Criteria:

* Non-reassuring fetal heart tracing, vaginal bleeding, chorioamnionitis or any indication for delivery at admission.
* Allergy to penicillin, erythromycin, or azithromycin.
* Multiple gestations.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Latency period | Number of days from PPROM to delivery, assessed up to 105 days
  Time from PPROM to delivery between the two treatments

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, MBA, Principal Investigator — Inova Health Care Services
Locations (2):
- United States (2):
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Eastern Viriginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navathe R, Schoen CN, Heidari P, Bachilova S, Ward A, Tepper J, Visintainer P, Hoffman MK, Smith S, Berghella V, Roman A. Azithromycin vs erythromycin for the management of preterm premature rupture of membranes. Am J Obstet Gynecol. 2019 Aug;221(2):144.e1-144.e8. doi: 10.1016/j.ajog.2019.03.009. Epub 2019 Mar 20. PMID 30904320
- [Background] Drassinower D, Friedman AM, Obican SG, Levin H, Gyamfi-Bannerman C. Prolonged latency of preterm prelabour rupture of membranes and neurodevelopmental outcomes: a secondary analysis. BJOG. 2016 Sep;123(10):1629-35. doi: 10.1111/1471-0528.14133. Epub 2016 May 31. PMID 27245741
- [Background] Prelabor Rupture of Membranes: ACOG Practice Bulletin, Number 217. Obstet Gynecol. 2020 Mar;135(3):e80-e97. doi: 10.1097/AOG.0000000000003700. PMID 32080050